CLINICAL TRIAL: NCT01744223
Title: A Phase 1/2 Dose Escalation Study Evaluating Safety and Feasibility of BPX-501 T Cells After Partially Mismatched, Related, T Cell-Depleted HSCT (Hematopoietic Stem Cell Transplant)
Brief Title: Safety Study of Gene Modified Donor T-cells Following Partially Mismatched Stem Cell Transplant
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bellicum Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BP-001
Expanded Access: NCT03639844 (No longer available)
Record Dates: First submitted 2012-12-05; First posted 2012-12-06 (Estimated); Last update posted 2022-07-12 (Actual); Status verified 2022-07

CONDITIONS: Acute Lymphoblastic Leukemia; Acute Myelogenous Leukemia; Lymphoma; Myelodysplastic Syndromes
Keywords: iCaspase9; iCasp9; Inducible Caspase; AP1903; Dimerizer drug; T depleted; Suicide gene; CD-34 selection; haplotransplantation; Graft versus host disease; Allogenic transplantation
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Lymphoma; Myelodysplastic Syndromes; Graft vs Host Disease | interventions — AP 1903 reagent

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- SCT, BPX-501 dose 1, Rimiducid if needed (Experimental): 2x10E5 BPX-501 (rivogenlecleucel) cells per kg infused after TCR alpha beta depleted donor stem cell transplant.
  Rimiducid: Dimerizer drug administered by intravenous infusion in those subjects with acute GVHD with no response to steroids and/or other aGVHD medications or worsening in stage or grade of aGVHD after 48 hours. Subjects with chronic GvHD who do not respond to steroids/systemic therapies within 7 days, or there is a worsening in cGVHD, patients may then receive rimiducid.
  Interventions: Biological: BPX-501 dose 1; Drug: Rimiducid; Procedure: SCT
- SCT, BPX-501 dose 2, Rimiducid if needed (Experimental): 5x10E5 BPX-501 (rivogenlecleucel) cells per kg infused after TCR alpha beta depleted donor stem cell transplant.
  Rimiducid: Dimerizer drug administered by intravenous infusion in those subjects with acute GVHD with no response to steroids and/or other aGVHD medications or worsening in stage or grade of aGVHD after 48 hours. Subjects with chronic GvHD who do not respond to steroids/systemic therapies within 7 days, or there is a worsening in cGVHD, patients may then receive rimiducid.
  Interventions: Drug: Rimiducid; Biological: BPX-501 dose 2; Procedure: SCT
- SCT, BPX-501 dose 3, Rimiducid if needed (Experimental): 1x10E6 BPX-501 (rivogenlecleucel) cells per kg infused after TCR alpha beta depleted donor stem cell transplant.
  Rimiducid: Dimerizer drug administered by intravenous infusion in those subjects with acute GVHD with no response to steroids and/or other aGVHD medications or worsening in stage or grade of aGVHD after 48 hours. Subjects with chronic GvHD who do not respond to steroids/systemic therapies within 7 days, or there is a worsening in cGVHD, patients may then receive rimiducid.
  Interventions: Drug: Rimiducid; Biological: BPX-501 dose 3; Procedure: SCT
- SCT, BPX-501 dose 4, Rimiducid if needed (Experimental): 3x10E6 BPX-501 (rivogenlecleucel) cells per kg infused after TCR alpha beta depleted donor stem cell transplant .
  Rimiducid: Dimerizer drug administered by intravenous infusion in those subjects with acute GVHD with no response to steroids and/or other aGVHD medications or worsening in stage or grade of aGVHD after 48 hours. Subjects with chronic GvHD who do not respond to steroids/systemic therapies within 7 days, or there is a worsening in cGVHD, patients may then receive rimiducid.
  Interventions: Drug: Rimiducid; Biological: BPX-501 dose 4; Procedure: SCT

INTERVENTIONS:
Biological: BPX-501 dose 1 — Subjects will receive 2x10E5 donor T cells/kg genetically modified with BPZ-1001 retroviral vector containing the iCasp suicide gene (BPX-501) after stem cell transplant.
  Other Names: rivogenlecleucel
  Arms: SCT, BPX-501 dose 1, Rimiducid if needed
Drug: Rimiducid — Dimerizer drug administered by intravenous infusion in those subjects who develop GVHD after infusion of BPX-501 cells.
  Other Names: AP1903
Biological: BPX-501 dose 2 — Subjects will receive 5x10E5 donor T cells/kg genetically modified with BPZ-1001 retroviral vector containing the iCasp suicide gene (BPX-501) after stem cell transplant.
  Other Names: rivogenlecleucel
  Arms: SCT, BPX-501 dose 2, Rimiducid if needed
Biological: BPX-501 dose 3 — Subjects will receive 1x10E6 donor T cells/kg genetically modified with BPZ-1001 retroviral vector containing the iCasp suicide gene (BPX-501) after stem cell transplant.
  Other Names: rivogenlecleucel
  Arms: SCT, BPX-501 dose 3, Rimiducid if needed
Biological: BPX-501 dose 4 — Subjects will receive 3x10E6 donor T cells/kg genetically modified with BPZ-1001 retroviral vector containing the iCasp suicide gene (BPX-501) after stem cell transplant.
  Other Names: rivogenlecleucel
  Arms: SCT, BPX-501 dose 4, Rimiducid if needed
Procedure: SCT — all subjects will receive an alpha beta depleted donor transplant as part of treatment

SUMMARY:
This study will evaluate patients with blood cell cancers who are going to have an allogeneic (donor) blood stem cell transplant from a partially matched relative. The research study will test whether immune cells, called T cells, which come from the donor relative and are specially grown in the laboratory and then given back to the patient along with the stem cell transplant (T cell addback), can help the immune system recover faster after the transplant. As a safety measure, these T cells have been "programmed" with a "self-destruct switch" so that if, after they have been given to the patient, the T cells start to react against the tissues (called "graft versus host" disease, GVHD), the T cells can be destroyed.

DETAILED DESCRIPTION:
This is a Phase1/2 dose escalation study evaluating the safety and feasibility of BPX-501 infused after partially mismatched, related (haploidentical), T cell-depleted HSCT. The purpose of this clinical trial is to determine whether BPX-501 infusion can facilitate engraftment, enhance immune reconstitution and potentially improve the graft versus leukemia (GVL) effect, with the potential for reducing the severity and duration of severe acute graft versus host disease (GvHD). The trial will evaluate the treatment of GvHD by the infusion of dimerizer drug (Rimiducid) in those subjects who present with GvHD that does not adequately respond to standard of care therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent
2. Age ≥ 18 years and ≤ 65 years
3. Deemed eligible for allogeneic stem cell transplantation
4. Lack of suitable conventional donor (i.e. 8/8 related or unrelated donor) or presence of rapidly progressive disease not permitting time to identify an unrelated donor
5. HLA typing will be performed at high resolution (allele level) for the HLA-A, -B, Cw, and DRBl, and loci

   * A minimum genotypic identical match of 4/8 is required.
   * The donor and recipient must be identical, as determined by high resolution typing, at least one allele of each of the following genetic loci: HLA-A, HLA-B, HLA-Cw, and HLA-DRB1
6. Subjects with adequate organ functions as measured by:

   1. Cardiac: Left ventricular ejection fraction at rest must be ≥ 45%
   2. Hepatic: Bilirubin ≤ 2.5 mg/dL and ALT, AST and Alkaline Phosphatase < 5 x ULN
   3. Renal: Serum creatinine within normal range for age or creatinine clearance, or with a recommended GFR ≥ 50 mL/min/1.73m2
   4. Pulmonary: FEV 1, FVC and DLCO (diffusion capacity) ≥ 50% predicted (corrected for hemoglobin); or O2 saturation > 92% on room air
7. Clinical diagnosis of one of the following:

   a. Acute Leukemia (includes T lymphoblastic lymphoma) in 2nd or subsequent complete remission (CR) i. Acute Lymphoblastic Leukemia (ALL) in 2nd or subsequent CR. ALL shall be morphologic remission at the time of transplant. Morphologic remission is defined that subjects with normal neutrophil and platelet counts, less than 5% blast cells in a bone marrow (BM) smear and no extramedullary disease ii. Acute Myeloid Leukemia (AML) in 2nd or subsequent CR with or without persistent minimal residual disease b. High-risk ALL in 1st CR (including features such as those in i-iii) i. Adverse cytogenetics such as t(9;22), t(1;19), t(4;11), MLL rearrangements ii. Subjects over 30 years of age, or iii. Time to complete remission was greater than 4 weeks. c. High-risk AML in 1st CR (including features such as those listed in i-vii) i. Greater than 1 cycle of induction therapy required to achieve remission ii. Preceding myelodysplastic syndrome (MDS) iii. Presence of FLT3 abnormalities iv. FAB M6 or M7 leukemia v. Adverse cytogenetics for overall survival such as those associated with MDS vi. Complex karyotype (>3 abnormalities), or vii. Any of the following: inv(3) or t(3;3), t(6;9), t(6;11), + 8 [alone or with other abnormalities except for t(8;21), t(9;11), inv(16) or t(16;16)], t(l1;19)(q23;p13.1) d. High risk Myelodysplastic Syndrome e. Non-Hodgkin's Lymphoma relapsed after autologous transplantation f. Non-Hodgkin's Lymphoma with insufficient autologous hematopoietic stem cells to undergo autologous transplantation g. CML i. in first chronic phase that has not attained at least a complete cytogenetic remission after exposure to at least 3 tyrosine kinase inhibitors ii. in accelerated phase that has not attained at least a complete cytogenetic remission iii. in second chronic phase
8. Performance status: Karnofsky score ≥60%.
9. Patient with hematologic malignancy not responding to /or not eligible for conventional therapy and are approved by Sponsor

Exclusion Criteria:

1. HLA 8/8 allele matched (HLA-A,-B,-Cw,-DRBl) related or unrelated donor able to donate.
2. Autologous hematopoietic stem cell transplant < 3 months prior to enrollment.
3. Pregnancy or breast-feeding.
4. Evidence of HIV infection or known HIV positive serology.
5. Current uncontrolled bacterial, viral or fungal infection (currently taking medication with evidence of progression of clinical symptoms or radiologic findings). The treating physician will make final determination.
6. Non-hematologic malignancy within prior three (3) years, with the exception of squamous cell or basal cell skin carcinoma.
7. Prior allogeneic hematopoietic stem cell transplant.
8. Subjects with a history of primary idiopathic myelofibrosis.
9. Bovine product allergy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2013-03 (Actual); Primary Completion 2019-10-09 (Actual); Study Completion 2032-10 (Estimated)

PRIMARY OUTCOMES:
BPX-501 Safety | 24 months
  To evaluate the safety of infusion of each of 4 dose cohorts of BPX-501 (2x105, 5x105, 1x106 and 3x106 cells/kg) after transplantation of partially mismatched T cell depleted hematopoietic stem cell transplant (HSCT)
Rimiducid Safety | 24 months
  To evaluate the safety of the infusion of the rimiducid in subjects who received BPX-501 and have developed visceral or steroid refractory graft-versus-host-disease
MTD | 24 months
  To determine the maximum dose of BPX-501 (up to 3x106 cells/kg) that results in an adjusted cumulative incidence by Day 100 of no more than 45% Grade II - IV aGVHD and / or no more than 17% Grade III -IV aGVHD.
Immune Reconstitution | 24 months
  To assess immune reconstitution for each dose cohort

SECONDARY OUTCOMES:
Efficacy- NRM | 100, 180 days and 1 year
  Non-Relapse Mortality (NRM)
Efficacy- DFS | 24 months
  Disease-free survival
Efficacy- TRM | 24 months
  Transplant related mortality (TRM)
Efficacy- Relapse | 24 months
  Incidence of Relapse
Incidence of engraftment | 24 months
  Evaluation of neutrophil and platelet engraftment, kinetics of donor cell engraftment and graft failure
GvHD | 24 months
  Incidence and severity of acute and chronic GvHD
GvHD post Rimiducid Administration | 24 months
  Time to resolution of acute GvHD after administration of Rimiducid
BPX-501 Safety Profile | 24 months
  Characterize the safety profile of BPX-501 including evaluation of high grade toxicity and infectious complications
Pharmacokinetics of Rimiducid | 24 months
  Pharmacokinetic disposition of Rimiducid

CONTACTS AND LOCATIONS:
Overall Officials: Bellicum Pharmaceuticals, Study Director — Bellicum Pharmaceuticals, Inc.
Locations (8):
- United States (8):
  - Emory University Winship Cancer Institute, Atlanta, Georgia
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Baylor Sammons Cancer Center, Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - Fred Hutchinson Cancer Research Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No